CLINICAL TRIAL: NCT03992898
Title: Establishment and Validation of Prognostic Nomograms for HBV-related Acute-on-Chronic Liver Failure in South of China
Brief Title: Nomogram Analysis for HBV Related Acute-on-chronic Liver Failure
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Bingliang, Clinical Professor, Sun Yat-sen University
Other Study IDs: Survival Study Cohort(SSC001)
Record Dates: First submitted 2019-06-19; First posted 2019-06-20 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic hepatitis cohort: In this cohort, patients were defined as type A acute-on-chronic liver failure (ACLF) patients who have chronic liver disease but without cirrhosis.
  Interventions: Other: No special intervention was suitable for this observational study
- Cirrhosis cohort: In this cohort, patients were defined as type B and type C ACLF patients with cirrhosis.
  Interventions: Other: No special intervention was suitable for this observational study

INTERVENTIONS:
Other: No special intervention was suitable for this observational study — Investegators divided patients into 3 corhort according to the liver condition at enrollment (i.e. chronic liver disease, compemsated cirrhosis, decompensated cirrhosis). All patients received standard medical treatment, including nutritional supplementation; administration of human serum albumin, fresh frozen plasma, antivirus treatment and appropriate treatment for complications. No special intervention was suitable for this observational study.

SUMMARY:
Acute-on-chronic liver failure (ACLF) is an acute deterioration of chronic liver diseases, which progresses rapidly, with a mortality rate of more than 50%.MELD score is used to evaluate the patients' condition. However, MELD score only concerned about the variables of total bilirubin, international normalize ratio (INR) and creatinine which is not enough to access ACLF patients' condition accurately.

Scholars of US and China suggested to divided ACLF patients into 3 subgroups base on the different "chronic liver disease" . Type A ACLF patients have chronic liver disease without cirrhosis. Type B ACLF patients with compensated cirrhosis, while type C ACLF patients with decompensated cirrhosis. Currently, no studies have assessed the prognosis of different types of ACLF patients, especially for HBV-related ACLF patients.

Investigators conducted a retrospective study which enrolls HBV-related ACLF patients between January 2010 and March 2018 in the Third Affiliated Hospital of Sun Yat-sen University. Clinical data, survival time and information regarding liver transplantation after enrolment were collected. A nomogram was formulated based on the results of multivariable Cox regression analysis. The performance of the nomogram was evaluated by the concordance index (C-index) and assessed by comparing nomogram-predicted vs observed Kaplan-Meier estimates of survival probability, and bootstraps with 1000 resamples were applied to these activities. Comparisons between the nomogram, MELD Score，MELD-Na Score and CTP Score in the entire population were performed and were tested by the C-index. A larger C-index indicated more accurate prognostic stratification.

DETAILED DESCRIPTION:
Acute-on-chronic liver failure (ACLF) is an acute deterioration of chronic liver diseases, which progresses rapidly, with a mortality rate of more than 50%. Liver transplantation is the only therapy that has been proven beneficial, but the number of liver donor is limited. MELD score is used to evaluate the patients' condition before transplantation to decide who is in greatest need. However, MELD score only concerned about the variables of total bilirubin, international normalize ratio (INR) and creatinine. Other important valuables such as age, hepatic encephalopathy, and indexes of infection (e.g. white blood cell counts) were excluded. Many studies showed that application of MELD score only is not enough to access the liver failure patients' condition accurately.

Both APASL and Chinese Society of Infectious Disease considered the "chronic liver disease" included chronic liver disease with/without cirrhosis. Scholars of US and China suggested to divided ACLF patients into 3 subgroups base on the different "chronic liver disease" . Type A ACLF patients have chronic liver disease without cirrhosis. Type B ACLF patients with compensated cirrhosis, while type C ACLF patients with decompensated cirrhosis. Currently, no studies have assessed the prognosis of different types of ACLF patients, especially for HBV-related ACLF patients.

Investigators conducted a retrospective study which enrolls HBV-related ACLF patients between January 2010 and March 2018 in the Third Affiliated Hospital of Sun Yat-sen University. Clinical data of demographic data, admission causes, cirrhosis complications, and precipitating events associated with acute decompensation or severe liver injury, laboratory measurements (e.g., serum albumin, sodium, alanine aminotransferase, aspartate aminotransferase, total bilirubin, INR and creatinine levels), mean arterial pressure, HBV infection biomarkers, HBV-DNA levels, antiviral treatment for HBV (nucleoside analogues, including lamivudine, adefovir, entecavir, telbivudine and tenofovir, within 6 months prior to and during hospitalisation), and prognosis would be collected. Survival time and information regarding liver transplantation after enrolment were also collected. A nomogram was formulated based on the results of multivariable Cox regression analysis. The performance of the nomogram was evaluated by the concordance index (C-index) and assessed by comparing nomogram-predicted vs observed Kaplan-Meier estimates of survival probability, and bootstraps with 1000 resamples were applied to these activities. Comparisons between the nomogram, MELD Score, MELD-Na Score and CTP Score in the entire population were performed and were tested by the C-index. A larger C-index indicated more accurate prognostic stratification.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years; Serum total bilirubin ≥ 10 mg/dl; International normalized ratio≥1.5 or prothrombin activity <40%; Complicated within 4 weeks by ascites and/or encephalopathy; Positive serum hepatitis B surface antigen for more than 6 months.

Exclusion Criteria:

* Drug induce liver diseases; Autoimmune liver diseases; Alcohol or drug abusers (average alcohol consumption >40g/d for men, >20g/d for women); Liver diseases caused by metabolic factors; Superinfection with hepatitis A, C, D, E viruses; Infected by HIV virus; Pregnancy or lactation; Liver failure caused by recurrence of hepatitis b after transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll a retrospective cohort of HBV related acute-on-chronic liver failure patients who were admitted to The Third affiliated Hospital of Sun Yat-sen University from January 2010 to March 2018.
Sampling Method: Probability Sample
Enrollment: 2739 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
survival status | 90 days
  Patients will be follow-up for 90 days until death or received liver transplantation. And survival days of each patients will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Bingliang Lin, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin B, Pan CQ, Xie D, Xie J, Xie S, Zhang X, Wu B, Lin C, Gao Z. Entecavir improves the outcome of acute-on-chronic liver failure due to the acute exacerbation of chronic hepatitis B. Hepatol Int. 2013 Jun;7(2):460-7. doi: 10.1007/s12072-012-9415-y. Epub 2013 Feb 11. PMID 26201778
- [Background] Duseja A, Choudhary NS, Gupta S, Dhiman RK, Chawla Y. APACHE II score is superior to SOFA, CTP and MELD in predicting the short-term mortality in patients with acute-on-chronic liver failure (ACLF). J Dig Dis. 2013 Sep;14(9):484-90. doi: 10.1111/1751-2980.12074. PMID 23692973
- [Background] Peng Y, Qi X, Tang S, Deng H, Li J, Ning Z, Dai J, Hou F, Zhao J, Wang R, Guo X. Child-Pugh, MELD, and ALBI scores for predicting the in-hospital mortality in cirrhotic patients with acute-on-chronic liver failure. Expert Rev Gastroenterol Hepatol. 2016 Aug;10(8):971-80. doi: 10.1080/17474124.2016.1177788. Epub 2016 Apr 25. PMID 27070325
- [Background] Moreau R, Jalan R, Gines P, Pavesi M, Angeli P, Cordoba J, Durand F, Gustot T, Saliba F, Domenicali M, Gerbes A, Wendon J, Alessandria C, Laleman W, Zeuzem S, Trebicka J, Bernardi M, Arroyo V; CANONIC Study Investigators of the EASL-CLIF Consortium. Acute-on-chronic liver failure is a distinct syndrome that develops in patients with acute decompensation of cirrhosis. Gastroenterology. 2013 Jun;144(7):1426-37, 1437.e1-9. doi: 10.1053/j.gastro.2013.02.042. Epub 2013 Mar 6. PMID 23474284
- [Background] Jalan R, Pavesi M, Saliba F, Amoros A, Fernandez J, Holland-Fischer P, Sawhney R, Mookerjee R, Caraceni P, Moreau R, Gines P, Durand F, Angeli P, Alessandria C, Laleman W, Trebicka J, Samuel D, Zeuzem S, Gustot T, Gerbes AL, Wendon J, Bernardi M, Arroyo V; CANONIC Study Investigators; EASL-CLIF Consortium. The CLIF Consortium Acute Decompensation score (CLIF-C ADs) for prognosis of hospitalised cirrhotic patients without acute-on-chronic liver failure. J Hepatol. 2015 Apr;62(4):831-40. doi: 10.1016/j.jhep.2014.11.012. Epub 2014 Nov 22. PMID 25463539
- [Background] Silva PE, Fayad L, Lazzarotto C, Ronsoni MF, Bazzo ML, Colombo BS, Dantas-Correa EB, Narciso-Schiavon JL, Schiavon LL. Single-centre validation of the EASL-CLIF consortium definition of acute-on-chronic liver failure and CLIF-SOFA for prediction of mortality in cirrhosis. Liver Int. 2015 May;35(5):1516-23. doi: 10.1111/liv.12597. Epub 2014 Jun 6. PMID 24840673
- [Background] Jalan R, Yurdaydin C, Bajaj JS, Acharya SK, Arroyo V, Lin HC, Gines P, Kim WR, Kamath PS; World Gastroenterology Organization Working Party. Toward an improved definition of acute-on-chronic liver failure. Gastroenterology. 2014 Jul;147(1):4-10. doi: 10.1053/j.gastro.2014.05.005. Epub 2014 May 20. No abstract available. PMID 24853409
- [Background] Luo Y, Xu Y, Li M, Xie Y, Gong G. A new multiparameter integrated MELD model for prognosis of HBV-related acute-on-chronic liver failure. Medicine (Baltimore). 2016 Aug;95(34):e4696. doi: 10.1097/MD.0000000000004696. PMID 27559979
- [Background] Shi KQ, Cai YJ, Lin Z, Dong JZ, Wu JM, Wang XD, Song M, Wang YQ, Chen YP. Development and validation of a prognostic nomogram for acute-on-chronic hepatitis B liver failure. J Gastroenterol Hepatol. 2017 Feb;32(2):497-505. doi: 10.1111/jgh.13502. PMID 27490495
- [Derived] Chen JF, Weng WZ, Huang M, Peng XH, Zhang J, Xiong J, He JR, Zhang SQ, Cao HJ, Gao B, Lin DN, Gao J, Gao ZL, Lin BL. The impact of serum thyroid-stimulation hormone levels on the outcome of hepatitis B virus related acute-on-chronic liver failure: an observational study. BMC Gastroenterol. 2022 Jul 7;22(1):330. doi: 10.1186/s12876-022-02406-7. PMID 35799116
- [Derived] Weng WZ, Chen JF, Peng XH, Huang M, Zhang J, Xiong J, Cao HJ, Lin BL. Risk factors for underlying comorbidities and complications in patients with hepatitis B virus-related acute-on-chronic liver failure. Epidemiol Infect. 2022 Jul 5;150:e147. doi: 10.1017/S0950268822001169. PMID 35788251
- [Derived] Chen JF, Weng WZ, Huang M, Peng XH, He JR, Zhang J, Xiong J, Zhang SQ, Cao HJ, Gao B, Lin DN, Gao J, Gao ZL, Lin BL. Derivation and Validation of a Nomogram for Predicting 90-Day Survival in Patients With HBV-Related Acute-on-Chronic Liver Failure. Front Med (Lausanne). 2021 Jun 16;8:692669. doi: 10.3389/fmed.2021.692669. eCollection 2021. PMID 34222294